CLINICAL TRIAL: NCT03166891
Title: Efficacy and Safety of Chiauranib in Relapsed/Refractory Ovarian Cancer: a Single-arm, Open-label, Multi-site, Exploratory Study
Brief Title: Phase Ib Study of Chiauranib in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR102
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer, relapsed or refractory,chiauranib
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — chiauranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chiauranib (Experimental): Patients take Chiauranib capsules 50mg, orally once daily, 28 days as a cycle.
  Interventions: Drug: Chiauranib

INTERVENTIONS:
Drug: Chiauranib — Take 50mg orally once daily
  Other Names: CS2164

SUMMARY:
Chiauranib may stop the growth of tumor cells by blocking Aurora kinase B（Aurora B）、VEGFR/PDGFR/c-Kit、CSF-1R targets. This clinical trial is studying the efficacy and safety of chiauranib(50mg，QD，PO) works in treating patients with relapsed or refractory ovarian cancer, in the meantime, exploring the latent biomarkers accompany with chiauranib, as well as the relevancy of which and clinical benefit.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety include adverse events, vital signs, laboratory tests ,etc., of Chiauranib in ovarian cancer patients due to the outcomes of the phase I study, and to explore the relevance between the latent biomarkers of Chiauranib and clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 yrs and ≤70 yrs;
2. Histological or cytological confirmation of epithelial ovarian cancer, carcinoma tubae, or primary peritoneal carcinoma.
3. Patients have received platinum containing chemotherapy, a) platinum resistant disease (disease progression within 6 months of the last receipt of platinum-based chemotherapy), the disease has progressed or relapsed after at least 2 different chemotherapy regimens; b) platinum sensitive disease (disease progression after 6 months of the last receipt of platinum-based chemotherapy), the disease has progressed or relapsed at least 2 different chemotherapy regimens, or the patients refuse any chemotherapy.
4. At least 1 lesion can be accurately measured, as defined by RECIST1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Subjects received anti-cancer therapy (including chemotherapy, radiotherapy, immunotherapy and surgical therapy, et al) should beyond 4 weeks prior to study entry; Subjects received mitomycin chemotherapy should beyond 6 weeks prior to study entry.
7. Laboratory criteria are as follows:

   Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.5×109/L ; platelets >=90×109/L Biochemistry test: total bilirubin≦1.5×ULN; alanine aminotransferase(ALT) ,aspartate aminotransferase(AST)≦1.5×ULN; (ALT,AST≦5×ULN if liver involved) ;serum creatinine(cr)≦1.5×ULN; Coagulation test: International Normalized Ratio (INR) < 1.5.
8. Life expectancy of at least 12 weeks.
9. Willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with prior invasive malignancies with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ, unless received curative treatment and with documented evidence of no recurrence in the past five years;
2. Clinical evidence of central nervous system involvement;
3. Have uncontrolled or significant cardiovascular disease, including:

   1. Congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months prior to study entry; arrhythmia, or Left Ventricular Ejection Fraction (LVEF) < 50% requiring treatment with agents during screening stage.
   2. primary cardiomyopathy(dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al)
   3. History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 470 ms prior to study entry
   4. Symptomatic coronary heart disease requiring treatment with agents
   5. Uncontrolled hypertension (> 140/90 mmHg) by single agent.
4. Have active bleeding current thrombotic disease, patients with bleeding potential ,or receiving anticoagulation therapy; within 2 months prior to screening;
5. Proteinuria positive(≥1g/24h).
6. History of deep vein thrombosis or pulmonary embolism;
7. Have unsolved toxicities (> grade 1) from prior anti-cancer therapy;
8. Have clinical significant gastrointestinal abnormality, e.g., unable to swallow, chronic diarrhea, ileus, that would impair the ingestion,transportation or absorption of oral agents, or patients undergone gastrectomy.
9. History of organ transplantation.
10. Major surgery within 6 weeks and minor surgery within 2 weeks prior to screening (excluding placement of vascular access or biopsy) that involved general anaesthesia or respiratory assistance.
11. Serologically positive for HIV, hepatitis B or C, or other serious infectious diseases.
12. History of interstitial lung disease(ILD).
13. Previous treatment with aurora kinase inhibitors.
14. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document or the operation and compliance of study;
15. Candidate with drug and alcohol abuse.
16. Participants of reproductive potential not willing to use adequate contraceptive measures for the duration of the study (both male and female participants).Pregnant or breastfeeding women. Female participants must have a negative urinary or serum pregnancy test when done or have evidence of post-menopausal status (Defined as absence of menstruation for greater than 12 months, bilateral oophorectomy or hysterectomy).
17. Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Overall response rate(ORR) | assessed up to 2 years
  ORR will be calculated from the data obtained from the end visit

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | measured through 2 years
  measured by adverse events (AE), serious adverse events (SAE), abnormal vital signs，electrocardiograph(ECG) and abnormal laboratory results according to CTCAE V4.03
Progression-free survival (PFS) | assessed up to 2 years
  From date of treatment until the date of first documented progression or date of death from any cause, whichever came first
Time to progression(TTP) | through treatment completion, up to 2 years
  duration from date of treatment until the date of first documented progression
Duration of response (DOR) | assessed up to 2 years
  From the first date of response until the date of first documented progression
Overall survival(OS) | assessed up to 2 years
  Time from treatment to death from any cause
16 week-disease control rate(16W-DCR) | assessed up to 2 years
  Rate of the patients with disease control longer than 6 weeks

OTHER OUTCOMES:
immunohistochemical(IHC) staining results of Aurora B、CSF-1R and Myc protein | assessed up to 2 years
  The IHC staining results were assigned a mean follows: 0, negative; 1, weak; 2, moderate; and 3, strong. The frequency of positive cells was defined as follows: 0, less than 5%; 1, 5% to 25%; 2, 26% to 50%; 3, 51% to 75%; and 4,greater than 75%.
Any single mutation of oncogene and copy number variation in ctDNA(single gene analysis) | assessed up to 2 years
Mutation of polygene and copy number variation in signal pathway(multi-gene analysis) | assessed up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li J, Liu J, Yin R, Zou D, Zheng H, Cao J, Chen Z, Sun W, Gao Y, Zhang S, Zeng L, An R, Lu X, Ye S, Wu X. Efficacy and safety of chiauranib in a combination therapy in platinum-resistant or refractory ovarian cancer: a multicenter, open-label, phase Ib and II study. Mol Cancer. 2024 Aug 9;23(1):162. doi: 10.1186/s12943-024-02076-x. PMID 39123210